CLINICAL TRIAL: NCT04498910
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of LY3451838 in Adults With Treatment-Resistant Migraine
Brief Title: A Study of LY3451838 in Participants With Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17124; J1H-MC-LAJB (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1500 milligrams (mg) LY3451838 (Experimental): Participants received a single intravenous (IV) dose of 1500 mg LY3451838.
  Interventions: Drug: LY3451838
- Placebo (Placebo Comparator): Participants received a single IV dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3451838 — Administered IV
  Arms: 1500 milligrams (mg) LY3451838
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The reason for this study is to see if the study drug LY3451838 is safe and effective in participants who have migraine that have not responded to other preventive treatments.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of migraine with a history of migraine headaches of at least 1 year prior, and migraine onset prior to age 50.
* Have completed at least 80% of required daily diary entries during the start of the study.
* Have documentation of previous failure of 2 to 4 standard-of-care migraine preventive medication categories in the past 10 years.
* Women of child-bearing potential must test negative for pregnancy as indicated by a negative serum pregnancy test and negative urine pregnancy test.
* Women of child-bearing potential who are abstinent or in a same sex relationship must agree to either remain abstinent or to avoid sexual relationships with males.
* Women of child-bearing potential who are not abstinent, must agree to use one highly effective method of contraception, or a combination of two effective methods of contraception during the study, as well as 5 months following.
* Women not of childbearing potential may participate and include those who are: A. Infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy or tubal ligation) or congenital anomaly; or B. Post-menopausal - defined as either:

  * i. a woman at least 40 years of age with an intact uterus, not on hormone therapy, who has cessation of menses for at least 1 year without an alternative medical cause, and a follicle-stimulating hormone greater than (>) 40 multi-international units per milliliter (mIU/mL); or
  * ii. a woman 55 or older not on hormone therapy, who has had at least 12 months of spontaneous amenorrhea; or
  * iii. a woman at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy

Exclusion Criteria:

* Are currently enrolled in any other clinical study or any other type of medical research judged not to be compatible with this study.
* Have participated, within the last 30 days or 5-half-lives (whichever is longer), in a clinical study involving any investigational product. If the half-life of the investigational product is unknown, 6 months should have passed prior.
* Known hypersensitivity or intolerance to monoclonal antibodies or other therapeutic proteins, or to common antihistamines, epinephrine, methyl prednisone or other systemic corticosteroids.
* Are currently receiving medication or other treatment for prevention of migraine headaches. Participants must have discontinued such medications or treatments at least 2 weeks prior. Botulinum toxin A or B that has been administered in the head or neck area use must be discontinued at least 3 months prior. Nerve blocks or device use (such as transcranial magnetic stimulation or electrical nerve stimulation) in the head or neck area for migraine treatment must be discontinued at least 30 days prior. Anti-calcitonin gene-related peptide (CGRP) antibodies must be discontinued at least 5 half-lives prior.
* Have previously failed more than 4 migraine preventive medication categories in the past 10 years due to inadequate efficacy (that is, maximum tolerated dose for at least 2 months) and/or safety / tolerability reasons.
* History of cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, retinal migraine, typical aura without headache, complications of migraine and migraine with brainstem aura (basilar-type migraine).
* In the 3 months prior, have other types of headache besides migraine, tension type headache, or medication overuse headache (MOH). (In other words, participants can have migraine, tension type headache, or MOH in the 3 months prior, but they cannot have other types of headache in that time).
* History of head or neck injury within last 6 months.
* History of traumatic cervical or head injury associated with significant change in the quality or frequency of headaches.
* Have reading of electrocardiogram (ECG) showing abnormalities considered incompatible with the study.
* Any liver tests outside the normal range.
* Evidence of significant active or unstable psychiatric disease.
* Women who are pregnant or nursing.
* Participants who have used opioids or barbiturate-containing analgesic >4 days per month for the treatment of pain in each of the past 3 months.
* History of drug or alcohol abuse/dependence within 1 year.
* Have a positive urine drug screen for illicit drugs.
* Are unwilling or unable to comply with the use of data collection devices.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - 21st Century Neurology, a division of Xenoscience, Phoenix, Arizona
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Renstar Medical Research, Ocala, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Bio Behavioral Health, Toms River, New Jersey
  - Health Research of Hampton Roads Inc, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Johnson MP, Krikke-Workel J, Patel CN, Morin SM, Turner PK, Clark KA, Donley D, Jin Y, Johnson KW, Vincent M, Stille JR, Broad LM, Patel A. Preclinical and clinical evaluation of LY3451838, a PACAP-neutralizing monoclonal antibody, in randomized, double-blind, placebo-controlled phase 1 and phase 2 studies involving healthy adults and adults with treatment-resistant migraine. Cephalalgia. 2025 Aug;45(8):3331024251368757. doi: 10.1177/03331024251368757. Epub 2025 Aug 21. PMID 40836866
- See also: A Study of LY3451838 in Participants With Migraine — https://trials.lilly.com/en-US/trial/283602

RESULTS

PARTICIPANT FLOW:
Groups:
- 1500 Milligram (mg) LY3451838: Participants received a single intravenous (IV) dose of 1500 mg LY3451838.
Period: Overall Study
Arm/Group | 1500 Milligram (mg) LY3451838 | Placebo
Started | 19 | 19
Received at Least One Dose of Study Drug | 19 | 19
Completed | 16 | 17
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 1500 mg LY3451838: Participants received a single IV dose of 1500 mg LY3451838.
- Total: Total of all reporting groups
Arm/Group | 1500 mg LY3451838 | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (10.84) | 48.0 (12.59) | 48.3 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 19 | 16 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 38
Monthly Number of Migraine Headache Days [Mean (Standard Deviation); unit: migraine days per month] — Migraine Headache Day is a calendar day on which a migraine or probable migraine occurs. Per International Headache Society [IHS] International Classification of Headache Disorders version 3 [ICHD-3], migraine is defined as a headache, with or without aura, of >=30 minutes duration with the following required features (A) At least 2 of the following headache characteristics: Unilateral location;Pulsatile quality;Moderate/severe pain intensity;Aggravation/causing avoidance of routine physical activity (B) During headache at least 1 of the following: Nausea/vomiting;Photophobia and phonophobia.
  migraine days per month | 14.0 (6.21) | 13.0 (7.71) | 13.5 (6.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Monthly Migraine Headache Days During 1-Month
Description: Migraine Headache Day is a calendar day on which a migraine or probable migraine headache occurs. Per International Headache Society [IHS] International Classification of Headache Disorders version 3 [ICHD-3], migraine is defined as a headache, with or without aura, of >=30 minutes duration with both of the following required features (A) At least 2 of the following headache characteristics: Unilateral location; Pulsatile quality; Moderate or severe pain intensity; Aggravation by or causing avoidance of routine physical activity (B) During headache at least 1 of the following: Nausea and/or vomiting; Photophobia and phonophobia. Least square mean was assessed using Bayesian Mixed Model Analysis with baseline number of monthly migraine headache days as a covariate.
Time Frame: Baseline, Month 1
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: migraine days per month
Arm/Group | 1500 mg LY3451838 | Placebo
Number analyzed (Participants) | 19 | 19
migraine days per month | -3.8 [-5.8 to -1.7] | -2.7 [-5.0 to -0.3]
Statistical Analysis 1: Comparison: 1500 mg LY3451838 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Difference in Estimated change = -1.1, 95% CI 2-sided [-3.6 to 1.2], Standard Error of Mean 1.2

2. Secondary Outcome: Change From Baseline in the Number of Monthly Headache Days During 3-Month
Description: as for outcome 1
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: migraine days per month
Arm/Group | 1500 mg LY3451838 | Placebo
Number analyzed (Participants) | 19 | 19
migraine days per month | -3.6 [-5.9 to -1.4] | -2.2 [-4.7 to 0.4]
Statistical Analysis 1: Comparison: 1500 mg LY3451838 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Difference in Estimated change = -1.5, 95% CI 2-sided [-4.2 to 1.0], Standard Error of Mean 1.3

3. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in Monthly Migraine Headache Days
Description: Percentage of Participants with ≥50% Reduction from Baseline in Monthly Migraine Headache Days are reported.
Time Frame: Month 1
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | 1500 mg LY3451838 | Placebo
Number analyzed (Participants) | 19 | 19
Percentage of participants | 21.1 | 26.3

4. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Events (TEAEs)
Description: Number of Participants with at least one TEAEs are reported. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to 5 Months
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1500 mg LY3451838 | Placebo
Number analyzed (Participants) | 19 | 19
Participants | 11 | 13

5. Secondary Outcome: Number of Participants With at Least One Serious Adverse Events (SAEs)
Description: Number of Participants with at least one SAEs are reported. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to 5 Months
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1500 mg LY3451838 | Placebo
Number analyzed (Participants) | 19 | 19
Participants | 1 | 0

6. Secondary Outcome: Pharmacokinetics (PK): Area Under the Serum Concentration-time Curve From Time 0 to the Last Measurable Serum Concentration (AUC 0-t) of LY3451838
Description: PK: AUC(0-t) of LY3451838
Time Frame: Pre-infusion, end of infusion, 3hours(h), 365h, 730h, 1095h, 1460h, 1825h, 2190h, 2920h, 3650h post-infusion
Population: All randomized participants who received at least one dose of LY3451838 and had evaluable serum concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg*h/mL)
Arm/Group | 1500 mg LY3451838
Number analyzed (Participants) | 19
microgram*hour per milliliter (μg*h/mL) | 176000 (26.5)

7. Secondary Outcome: PK: Maximum Observed Serum Concentration (Cmax) of LY3451838
Description: PK: Cmax of LY3451838
Time Frame: Pre-infusion, end of infusion, 3hours(h), 365h, 730h, 1095h, 1460h, 1825h, 2190h, 2920h, 3650h post-infusion
Population: All randomized participants who received at least one dose of LY3451838 and had evaluable serum concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/ml)
Arm/Group | 1500 mg LY3451838
Number analyzed (Participants) | 19
microgram per milliliter (µg/ml) | 613 (32.6)

ADVERSE EVENTS:
Time Frame: Baseline up to 5 Months
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 1500 mg LY3451838 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 14/19 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1500 mg LY3451838 (N=19) | Placebo (N=19)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1500 mg LY3451838 (N=19) | Placebo (N=19)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 4 (5) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase abnormal (Investigations) | 0 (0) | 1 (1)
Biopsy breast normal (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Lumbar puncture (Investigations) | 1 (1) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Aura (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/18 (0) | 1/18 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT04498910/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT04498910/SAP_001.pdf